CLINICAL TRIAL: NCT00391820
Title: A Phase II, Randomized, Double-Blind, Placebo-Controlled Study of TD-5108 for the Treatment of Chronic Constipation
Brief Title: Evaluate the Safety and Efficacy of a 5-HT4 Agonist in Chronic Constipation (ACCORD Trial)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alfasigma S.p.A. (Industry)
Collaborators: Theravance Biopharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0038
Record Dates: First submitted 2006-10-20; First posted 2006-10-24 (Estimated); Last update posted 2025-07-08 (Actual); Status verified 2014-12

CONDITIONS: Chronic Constipation
Keywords: constipation; chronic; bowel function
MeSH Terms: conditions — Constipation; Bronchiolitis Obliterans Syndrome | interventions — TD-5108

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: TD-5108

SUMMARY:
Study 0038 compares the safety and effectiveness of an investigational drug, TD-5108 with placebo (a sugar pill) for the treatment of chronic constipation.

ELIGIBILITY:
Inclusion Criteria:

* Meet ROME III Criteria

Exclusion Criteria:

* Constipation caused by:colonic etiology, pelvic floor dysfunction, metabolic disturbances, neurologic disturbances,concomitant medications affecting bowel function
* Chronic treatment with anticholinergics, narcotic analgesics
* Irritable Bowel Syndrome

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 360 (Estimated)
Dates: Start 2006-10; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
- Clinical response

CONTACTS AND LOCATIONS:
Locations (1):
- Breco Research, Houston, Texas, United States

REFERENCES:
- [Derived] Goldberg M, Li YP, Johanson JF, Mangel AW, Kitt M, Beattie DT, Kersey K, Daniels O. Clinical trial: the efficacy and tolerability of velusetrag, a selective 5-HT4 agonist with high intrinsic activity, in chronic idiopathic constipation - a 4-week, randomized, double-blind, placebo-controlled, dose-response study. Aliment Pharmacol Ther. 2010 Nov;32(9):1102-12. doi: 10.1111/j.1365-2036.2010.04456.x. Epub 2010 Sep 22. PMID 21039672